CLINICAL TRIAL: NCT04244123
Title: Application of Web-based Adherence Information Integrated Nurse-led Monitoring Clinic for Growth Hormone Treatment in Children
Brief Title: Web-based Adherence Information Integrated Nurse-led Monitoring Clinic
Acronym: WAIN-MC
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00672
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Short Stature; Growth Hormone Treatment
Keywords: Growth Hormone
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- growth hormone deficiency: growth hormone deficiency, requiring growth hormone treatment
  Interventions: Combination Product: integrated information and nurse led telephone clinic
- small for gestational age: small for gestational age and failure of post natal catch up height gain, requiring growth hormone treatment
  Interventions: Combination Product: integrated information and nurse led telephone clinic
- Turner syndrome: short stature due to Turner syndrome, on growth hormone treatment
  Interventions: Combination Product: integrated information and nurse led telephone clinic
- chronic renal failure: short stature due to chronic renal failure, treated with growth hormone treatment
  Interventions: Combination Product: integrated information and nurse led telephone clinic
- Prader Willi syndrome: short stature due to Prader Willi syndrome, treated with growth hormone treatment
  Interventions: Combination Product: integrated information and nurse led telephone clinic

INTERVENTIONS:
Combination Product: integrated information and nurse led telephone clinic — combining web-based information from easypod connect with nurse led telephone clinic

SUMMARY:
Non-adherence is a recognized problem with growth hormone treatment in children. In this study, we aim to utilize web-based information derived from easypod growth hormone injection devices and easypod connect devices in a nurse-led telephone clinic to improve adherence and therefore optimize growth. Our primary aim is to test height SDS change over a 12 month period. Our secondary aims are to test adherence, acceptance/satisfaction and qualitative assessment.

DETAILED DESCRIPTION:
Background:

Recombinant human growth hormone (GH) is used in the treatment of short stature due to growth hormone deficiency, Turner syndrome, Prader Willi syndrome, small for gestational age with failure of catch up growth, chronic renal failure and SHOX deficiency. Growth hormone is administered at home as daily injections and given over several years. Administration of growth hormone involves considerable commitment from parents and families and incurs significant cost to the NHS in the UK. Current treatment regimens using a range of GH formulations are not based on drug efficacy, cost effectiveness or cost of treatment.

It is well recognised that adherence to treatment is directly correlated to height performance in patients receiving GH. Several studies have indicated better height outcomes through use of technology to enhance patient adherence. The standard model of care of GH therapy involves patients returning to review appointments with clinicians for GH monitoring and dose adjustment. This model requires travel to hospitals at regular intervals (3-4 monthly), causing disruption to regular routines, inconveniencing family commitments, education and school. Importantly, this model does not encourage adherence or compliance with GH and relies on individual patient and family initiative to ensure treatment delivery. Alternative and more user-friendly models of care promoting greater adherence to GH are required to improve efficiency of GH treatment outcomes.

We have proposed a novel model of GH treatment monitoring integrating web-based adherence information in paediatric endocrine specialist nurse-led telephone clinics. A specialist nurse-led telephone clinic for management of growth hormone already exists at the Royal Manchester Children's Hospital (RMCH) and generates positive feedback from parents and families whilst releasing capacity in face to face growth clinics. The WAIN-MC model integrates and improves this specialist nurse-led clinic with web-based GH adherence information as a clinical innovation. The proposed model enables remote monitoring without travel to the hospital, review of growth performance in relation to adherence information and improved engagement of parents/families, thereby increasing adherence, satisfaction and height gain.

Rationale:

Current models of GH treatment are not targeted towards increasing adherence and achieving improved height gain. It is important to explore alternative models of care using GH that improve adherence to treatment and result in improved height outcome whilst enhancing patient satisfaction. The WAIN-MC model represents a clinical innovation which requires testing for utility in a pilot study prior to wider application in the NHS.

The WAIN-MC feasibility study provides an alternative treatment model that might improve adherence of treatment, resulting in greater height outcome than with the current standard model of hospital review. This study is based on a telephone clinic run by specialist nurses who are able to access information about treatment adherence through easypod connect. This model enables greater understanding of adherence patterns correlated to height gain without requiring additional hospital reviews and the stress of frequent visits to the hospital. It is likely to be better accepted by parents and families, thereby fostering greater adherence and culminating in greater efficiency of treatment. WAIN-MC represents the application of digital technology in the achievement of improved treatment outcomes in children receiving GH treatment.

Previous findings and data from other studies It is well recognised that an important component of treatment outcome with GH is adherence. However, non-adherence is common among children and families receiving treatment with height outcomes being limited by and correlated with the degree of non-adherence [1]. In spite of efforts made by healthcare professionals, long term adherence with GH treatment is suboptimal and widespread [2], with one study reporting 30% good adherence [3].

Several devices are available to inject or transject GH for treatment in children. Only one device records the number of the injections and the efficiency of dose injection administered - Saizen easypod™ manufactured by Merck Healthcare KGaA. Easypod can also dock into a 4G connected device, easypod connect™ which uploads adherence as digital information specific to the patient. A recent study showed good adherence using easypod connect with the magnitude of 2 year catch-up height gain correlated to high adherence levels [4]. In the multi-centred longitudinal observational study (ECOS study) involving 1190 patients, median adherence with GH treatment was high at 93.7% in the first year [5]. However, adherence decreased with increasing treatment duration with adherence rates progressively declining to 87.2% at 3 years, 75.5% at 4 years and 70.2% at 5 years. Thus the use of easypod GH and easypod connect is strongly associated with good adherence with GH treatment but is unable to prevent the reduction of adherence rates over longer durations of treatment.

The WAIN-MC clinical innovation integrates easypod connect with the structure of a specialist nurse-led telephone clinic for additive treatment outcome benefits for each component. It is expected that the synthesis model will not only reinforce adherence but also sustain this through regular clinical contact. WAIN-MC is a novel development and therefore has not been investigated for efficacy.

The following are the likely benefits of WAIN-MC to participants:

1. Improved height gain over 1 year of treatment; initial height gain is likely to correlate with optimal final height gain at the end of treatment
2. Improved patient and family satisfaction with WAIN-MC, reinforcing further adherence
3. Increased clinic capacity for standard clinic reviews
4. Improved cost efficiency of treatment with favourable financial cost of height gain and favourable total cost of treatment
5. Serve as a template for future studies in GH treatment and other forms of daily injectable therapy

Hypothesis:

We hypothesize the following:

1. The WAIN-MC model is a feasible option in the treatment of children with GH.
2. Adherence will improve by 10% from the time of entry to the study to the time at the end of the study.
3. Children on GH will gain 0.5 SD or more within one year of adopting WAIN-MC
4. Parents and families will find the application of WAIN-MC to their satisfaction and therefore provide positive qualitative feedback.

Objectives:

The study aims to investigate the utility of a nurse led clinic using easypod connect web-based GH adherence information in a one year feasibility study. The study will investigate if adherence with easypod GH improves by combining easypod connect with nurse led telephone monitoring clinics. The study will also investigate potential improvement in height gain over 12 months whilst adopting WAIN-MC.

Study design:

This is a feasibility study designed to investigate whether the WAIN-MC model is practical for use in this population. At present there are 70 patients enrolled on this model, which is a reasonable sample size to assess variation in auxology outcomes. Taking alpha as 0.05, and 90% power, a sample size of 70 will detect an effect size of 0.41, allowing for 10% dropout.

For the semi-structured interviews not all parents will consent and financial and time practicalities also constrain the sample size. All 70 patients will be invited to consent and a random selection of 15 individuals will be selected from those consenting to take part in a semi structured interview for feedback.

There are no controls groups for this feasibility study. Each patient will serve as his/her own control with comparison of adherence and auxology data between initial and final visits.

Study Design:

1. Patients All patients who receive easypod GH of age 1-14 years will be approached for consent to participate in the study. Patients may have any valid cause for short stature. These may include children with isolated growth hormone deficiency, multiple pituitary hormone deficiencies, and non-growth hormone deficient conditions such as small for gestational age with postnatal failure of height gain, chronic renal failure and Turner syndrome. Patients will be recruited to the study irrespective of diagnosis and will not be stratified by diagnosis at entry to the study. However, in analysis of data, subgroup analysis may be performed on groups such as those with isolated growth hormone deficiency, dependent on the frequency of recruitment.

   All patients will be identified at the start of the study. A one month period will be considered before the study commences to contact families for potential recruitment. Each patient will remain in the study for 12 months. The active study duration will be 18 months whereby all eligible patients will be recruited and followed up for a 12 month period. This period will be followed by a buffer period to gather necessary data for analysis. The timeline of the study is provided in the in Appendix 1
2. Procedures Health Research Authority/Ethical (IRAS 264053) and MFT approval will be achieved for this study prior to any study procedures commencing. Information for consent will be provided to the parents of patients eligible to participate in the study at study initiation.

Paediatric endocrine specialist nurse led face to face appointments at outpatients in RMCH will be set up on 3 days for explanation and patient recruitment. The appointments will be led by specialist nurses Sister Julie Jones and Sister Helen Pimlott and overseen by Dr I Banerjee, CI for the study. Dr Banerjee will undertake consent for this study from parents and carers.

Standard clinic reviews with hospital visits will continue in parallel. Investigations, dose changes and other treatment alterations will be continued as part of routine clinical care.

At the initial visit, the following information will be obtained:

1. Adherence information based on easypod connect data over the month previous to study entry will be recorded in the clinical research form (CRF). A hard copy of a screen capture image will be stored in the CRF for each patient.
2. Height will be measured by a Harpenden stadiometer at outpatients department in RMCH. Weight will be measured at the time using weighing scales. Information on age, sex, height and weight will be entered into the CRF. Puberty will not be assessed but information on puberty will be obtained from the previous or closest clinic review correspondence. Auxology (height, weight) will be converted to standard deviation scores using both UK 1990 centiles and WHO reference standards.
3. The educational qualifications of one or both parents will be noted using the International Standard Classification of Education (ISCED) 2011 [http://www.uis.unesco.org/Education/Documents/isced-2011-operational-manual.pdf]. The following categories will be used: 0 pre-primary education, 1 primary education, 2 lower secondary education, 3 upper secondary education, 4 post-secondary non-tertiary education, 5 short-cycle tertiary education, 6 Bachelor or equivalent, 7 Master or equivalent, 8 Doctoral or equivalent.

Following the initial visit, two nurse led telephone monitoring clinics will be set up at 4 and 8 months. Patients and families will be offered a choice of 3 days for each of the 4 and 8 month telephone clinic appointments. Each appointment will last for 20 minutes. The telephone appointment will be structured in the following format:

1. Ascertain dose of easypod GH, cartridge size of easypod GH and check if supplies are adequate.
2. Record special circumstances potentially influencing adherence.
3. Parent/carer reported adverse events
4. Obtain recent height and weight data from GP surgery measurements
5. Record advice regarding method of administration, needle size and depth of injection
6. Record parent perceptions of adherence and comparison with easypod connect information over previous 3 months.

A final face to face nurse led clinic review will be undertaken at outpatients in RMCH. Patients and families will be offered a choice of 3 days for the final study visit. At the final appointment, the following information will be obtained:

1. Auxology data
2. Adherence data over previous 3 months
3. Adverse events, if any
4. The highest education status will be re-ascertained in as per the International Standard Classification of Education (ISCED)] as stated at the initial visit.

A randomly chosen subset (n=15) will be invited to a semi structured interview to provide feedback. The interview will be conducted by Dr Jacqueline Nicholson, clinical psychologist at RMCH. The interview will last 30 minutes and will focus on:

1. A 5 point Likert scale of parent perception of satisfaction for WAIN-MC
2. A 5 point Likert scale of parent perception of preference for WAIN-MC as a future clinical model
3. Qualitative comments of suitability of WAIN-MC to patient care and suggestions for improvement

(3) Analysis

All variables will be explored to understand their form and completeness using appropriate descriptive statistics (N [%], mean [standard deviation] or median [interquartile range]) and graphics. No imputation will take place for missing data, but consideration may be made in the analyses in the event of large numbers.

The difference in height SDS between entry and final visit will be assessed by paired t-tests or non-parametric equivalent as appropriate.

Adherence data will be available on a daily basis, but for the main purposes of analysis will be reported as a percentage for each month (1-12). Trends in non-adherence on a daily basis will be explored graphically with consideration for recorded information, e.g. consecutive non adherence due to technical fault or missing doses due to illness or being away on holiday. Adherence data over a 12 month period will be collated into units of time, i.e. weeks or months and presented descriptively, with the aid of longitudinal graphs. If indicated longitudinal models will be used to describe any trends.

The difference in adherence at entry to the study (month 1) and final visit (month 12) will be tested by paired t-tests or non-parametric equivalent. The change will also be explored using multivariable regression models to adjust for age, sex, diagnosis and ISCED group. Univariate and multivariable linear regression model will be used to investigate the effect of adherence on height SDS, adjusting for age, sex, diagnosis and ISCED group.

Qualitative analysis Results from the patent satisfaction and patient preference questionnaires will be presented descriptively. Interviews will be transcribed verbatim and the six stages of Thematic Analysis will be used to analyse the interview data.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive easypod GH of age 1-14 years will be approached for consent to participate in the study. Patients may have any valid cause for short stature. These may include children with
* isolated growth hormone deficiency
* multiple pituitary hormone deficiencies
* non-growth hormone deficient conditions such as
* Small for gestational age with postnatal failure of height gain
* chronic renal failure and
* Turner syndrome. Patients will be recruited to the study irrespective of diagnosis and will not be stratified by diagnosis at entry to the study. However, in analysis of data, subgroup analysis may be performed on groups such as those with isolated growth hormone deficiency, dependent on the frequency of recruitment.

All patients will be identified at the start of the study. A one month period will be considered before the study commences to contact families for potential recruitment. Each patient will remain in the study for 12 months. The active study duration will be 18 months whereby all eligible patients will be recruited and followed up for a 12 month period. This period will be followed by a buffer period to gather necessary data for analysis.

Exclusion Criteria:

* Patients on growth hormone treatment but using other growth hormone devices Patients who are younger or older than the age limits.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with short stature, due to various causes and receiving growth hormone treatment as per licensed indications will be eligible for recruitment if they use the easypod growth hormone device.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
change in height SDS | 12 months
  difference in height SDS

SECONDARY OUTCOMES:
Adherence to medication | 12 months
  Percentage of Adherence to medication
Qualitative assessment | 12 months
  Semi structured interview to qualitatively assess family perspectives

OTHER OUTCOMES:
Family feedback | 12 months
  feedback regarding acceptance/satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Indi Banerjee, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Indraneel Banerjee, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
overall high level data to be shared but not patient identifiable information